CLINICAL TRIAL: NCT03936179
Title: Phase II Trial of High Dose PET/CT-guided Radiation Therapy With Concurrent Weekly Carboplatin and Paclitaxel in Localregionally Advanced Esophageal Cancer
Brief Title: High Dose PET/CT-guided Intensity Modulated Radiotherapy and Concurrent Chemotherapy in Esophageal Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Chen tingfeng, director,department of radiation therapy, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGH201921
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- high dose radiochemotherapy (Experimental): A total dose of 86 Gy to residual metabolic disease with concurrent chemotherapy
  Interventions: Radiation: high dose radiation therapy with concurrent chemotherapy

INTERVENTIONS:
Radiation: high dose radiation therapy with concurrent chemotherapy — standard dose of 50 Gy concurrent weekly with paclitaxel (45 mg/m2) and carboplatin (area under curve 1.5 ), immediately followed by hyperfractionated radiotherapy boost of 36 Gy in 30 fractions of 1.2 Gy to residual metabolic disease as defined by PET/CT

SUMMARY:
To assess the efficacy and feasibility of high-dose intensity-modulated radiotherapy with concurrent weekly paclitaxel and cisplatin for patients with locaregionally esophageal cancer

DETAILED DESCRIPTION:
Standard dose chemoradiotherapy (SCRT) results in poor local control for localregionally advanced esopgageal cancer patients. Most local failures occur in the gross tumor volume.[F-18]-fluorodeoxyglucose (FDG) PET/CT can identify residual metabolic disease (RMD). Hyperfractionated radiotherapy allows for delivering a higher dose without increasing late toxicity. Our previous phase I radiation dose escalation trial demonstrated that 86 Gy could be safely delivered to the RMD with concurrent weekly paclitaxel and cisplatin in advanced esophageal cancer.The aim of this phase II study is to examine the efficacy of this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have FDG-avid and histologically or cytologically proven esophageal cancer.
* Patients must be deemed unresectable disease or patient is not deemed operable due to medical reasons.
* Eastern Cooperative Oncology Group （ECOG） performance status 0 to 2 No prior radiation to the thorax that would overlap with the current treatment field.
* Patients with nodal involvement are eligible
* Adequate bone marrow, renal and hepatic functions as assessed by the following: Hemoglobin >/= 10.0 g/dl, Platelet count >/= 1 00,000/ mm^3,absolute granulocyte count (AGC) ≥2 × 10^9 cells/L,bilirubin and Aspartate transaminase ≤1.5 ×upper limit of normal (ULN), Creatinine </ =1 .5 times ULN.
* A signed informed consent must be obtained prior to therapy.
* No prior radiation to the thorax that would overlap with the current treatment field.

Induction chemotherapy is allowed.

Exclusion Criteria:

* The presence of a fistula.
* Prior radiotherapy that would overlap the radiation fields.
* gastroesophageal junction cancer or the lower third esophageal cancer invading the gastric wall.
* Uncontrolled concurrent illness including, but not limited to: Chronic Obstructive Pulmonary Disease(COPD) exacerbation or other respiratory illness, serious uncontrolled infection, symptomatic congestive heart failure (CHF),unstable angina pectoris, uncontrolled hypertension,or psychiatric illness/social situations that would limit compliance with the study requirements.
* Known hypersensitivity to paclitaxel.
* Any other condition or circumstance that would, in the opinion of the Investigator, make the patient unsuitable for participation in the study.
* Acquired Immune Deficiency Syndrome.
* Conditions precluding medical follow-up and protocol compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
overall survival rate | one year
  survival time was measured from the date of study enrollment to the date of death or last follow-up

SECONDARY OUTCOMES:
acute and late toxicities | 1 year
  Acute toxicities were graded according to the National Cancer Institute-Common Toxicity Criteria (NCI-CTC) version 4

CONTACTS AND LOCATIONS:
Overall Officials: Tingfeng Chen, MD, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No